CLINICAL TRIAL: NCT04885387
Title: X-ray-free Protocol for Pectus Deformities Based on Magnetic Resonance 1 Imaging and a Low-cost Portable Three-dimensional Scanning Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Ballouhey Xray
Record Dates: First submitted 2021-05-09; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-03

CONDITIONS: Pectus Deformity
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard protocol using chest CT (Other)
  Interventions: Device: chest CT
- Magnetic Resonance Imaging and a low-cost portable three-dimensional scanning device (Experimental)
  Interventions: Device: Magnetic Resonance Imaging and a low-cost portable three-dimensional scanning device

INTERVENTIONS:
Device: chest CT — chest CT pectus deformities diagnostic
  Arms: Standard protocol using chest CT
Device: Magnetic Resonance Imaging and a low-cost portable three-dimensional scanning device — Magnetic Resonance Imaging and a low-cost portable three-dimensional scanning device pectus deformities diagnostic
  Arms: Magnetic Resonance Imaging and a low-cost portable three-dimensional scanning device

SUMMARY:
Pectus excavatum (PE) and pectus carinatum (PC) are the most frequent chest wall deformities in humans. They are usually clinically recognized in early childhood or adolescence, with aggravation during the pubertal growth spurt. PE is a depression of the anterior chest wall, most frequently involving the lower sternum.

In this study we use simultaneously compared chest CT, MRI, and 3D scanning fro both PE and PC assessment .

The aim of this study is to compare a standard protocol using chest CT to a non-irradiant protocol with 3D scanning and MRI.

The primary endpoint was to assess the inter observer concordance and the correlation between the HI (Haller Index) evaluated with MRI and the EHI (External Haller index) evaluated with 3D scanning. The secondary endpoints were to assess the concordance with chest CT the variation of the HI evaluated in inspiration and expiration with MRI and also the correction index (CI) between chest CT and MRI in the PE group, .

ELIGIBILITY:
Inclusion Criteria:

* children (< 18 years of age)
* with a pectus deformity
* recent (within the past month) chest CT, cardiothoracic MRI, and 3D scanning data were available.

Exclusion Criteria:

-

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
To compare a standard protocol using chest CT to a non-irradiant protocol involving a low-cost portable three-dimensional scanner and MRI for all pectus deformities based on the Haller index (HI) | At 12 month

SECONDARY OUTCOMES:
To compare the Haller Index measured with CT and the HI measured with low-cost portable three-dimensional scanner | At 12 month
To compare the Haller Index measured with CT and the HI measured with MRI | At 12 month

CONTACTS AND LOCATIONS:
Locations (1):
- Service de chirurgie infantile, Limoges, France